CLINICAL TRIAL: NCT02830815
Title: Comparative Effects of Two Anesthetic Techniques on Auditory Brain Response in Children
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-8186
Record Dates: First submitted 2016-06-29; First posted 2016-07-13 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Auditory Brainstem Response
Keywords: Broadband click stimulus testing; General Anesthesia; Sevoflurane; Propofol; Amplitude latency; Wave V

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This will be a prospective, blinded, cross-over study to compare the effects of two anesthetic techniques on the interpretability of auditory brainstem response testing in children.

DETAILED DESCRIPTION:
The proposed study will be a single-center, prospective, crossover-controlled study of the two anesthetic techniques (propofol and sevoflurane). The investigators plan to enroll 80 patients who receive general anesthesia at Cincinnati Children's Hospital Medical Center Department of Radiology for ABR testing. A sample size recalculation will be performed during the study to determine the exact number of subjects necessary for sufficient power. As per standard anesthesia practice for this test in radiology department, all subjects will serve as their own control, receiving both anesthetic techniques within the same ABR testing session. The audiologist will employ broadband click stimulus testing after induction with Sevoflurane, after which the patient will be switched over to a propofol infusion and the sevoflurane stopped. After the completion of the remainder of the ABR (tone-burst testing), the audiologist will repeat the broadband click testing (now while under propofol anesthesia), and the results will be recorded. At this point, results will be de-identified, with the exception of which ear was tested and the intensity level, and these results will be reviewed by a panel of 5 audiologists. These audiologists will be blinded to the anesthetic technique and patient information. They will provide a judgment at each intensity level, for each ear whether or not a response is present (in a Yes/No format). A study coordinator blinded to the anesthetic technique will record the outcome data. The anesthesia providers and nursing team will not be blinded.

ELIGIBILITY:
Inclusion Criteria:

* 0 - 18 years old
* ASA status I, II, or III
* Scheduled for ABR with general anesthesia

Exclusion Criteria:

* Contraindication to sevoflurane or propofol
* ASA >3

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients will be recruited from the radiology ABR schedule
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-06; Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

PRIMARY OUTCOMES:
Qualitative interpretability of ABR testing in the same patient undergoing two anesthetic techniques | Participants will be followed for the duration of the ABR test approximately 60 - 90 minutes
  This will be measured by a blinded panel of audiologist review the two ABR click test results and provide judgment at each intensity level, for each ear and whether or not a response is present.

SECONDARY OUTCOMES:
Amplitude of Wave V of the ABR after broadband click stimulus | Participants will be followed for the duration of the ABR test approximately 60 - 90 minutes
Latency of Wave V of the ABR after broadband click stimulus | Participants will be followed for the duration of the ABR test approximately 60 - 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ali Kandil, DO, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kandil AI, Ok MS, Baroch KA, Subramanyam R, Mahmoud MA, McAuliffe JJ 3rd. Why a Propofol Infusion Should Be the Anesthetic of Choice for Auditory Brainstem Response Testing in Children. Anesth Analg. 2022 Apr 1;134(4):802-809. doi: 10.1213/ANE.0000000000005693. PMID 35113042